CLINICAL TRIAL: NCT05835791
Title: Prospective Cohort for the sEcoNDary Prevention of Ventricular Tachycardia in Patients With Cardiomyopathies (END-VT) Study
Brief Title: END - VT Cohort Study
Acronym: END VT
Status: Recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Maritime Heart Centre (Other)
Responsible Party: Sponsor
Other Study IDs: SAPP0013
Record Dates: First submitted 2023-04-06; First posted 2023-04-28 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Ventricular Tachycardia; Implantable Defibrillator User; ICD
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ventricular tachycardia (VT) is a life-threatening cardiac rhythm disturbance which leads to sudden cardiac death (SCD), ventricular fibrillation, electrical storm, hemodynamic collapse, and syncope. VT patients with cardiomyopathy (diseased/scarred cardiac muscle) have the highest risk of SCD (<1-4%) and recurrent VTs (15-35%). Although an implantable cardiac defibrillator (ICD) is the most effective treatment option to prevent SCD, it does not eliminate it. Without VT prevention, recurrent VT and ICD shocks may increase the risk of heart failure and death.

The primary objective is to determine the optimal treatment strategy to maximize event-free survival among cardiomyopathy patients with ventricular tachycardia (VT) by the creation of a prospective, multicenter, longitudinal cohort. Also, the investigators will evaluate the epidemiology of VT, adherence to guidelines, safety, effectiveness, and cost-effectiveness of current treatment options for secondary prevention of VT in the real-world Canadian VT population.

DETAILED DESCRIPTION:
The END-VT study is a multicenter, prospective, longitudinal real-world cohort study of patients with cardiomyopathy-related VT. Patients with ischemic and non-ischemic cardiomyopathy are followed from their first VT event till at least 3 years of follow-up or death, whichever is first. Outcomes of VT events are captured by ICD remote monitoring and are adjudicated by experienced clinical investigators blinded to the center and treatments. The primary objective of END-VT is to determine the optimal treatment strategy to maximize event-free survival among cardiomyopathy patients with VT. The investigator will also assess the real-world burden of disease, treatment challenges, adherence to guidelines, sex differences, and safety, effectiveness, and cost-effectiveness of VT treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Documented sustained ventricular arrhythmia (>30 seconds as documented by an ECG, cardiac monitor, AED, and/or intracardiac pacemaker/ICD electrograms (EGMs);
2. First (new) diagnosis of VT;
3. Presence of or plan for ICD implant during index hospitalization;
4. Diagnosis of cardiomyopathy (ie. ICM, hypertrophic, dilated, restrictive, arrhythmogenic cardiomyopathy, or other scar),
5. ICD clinic follow-up planned, and
6. Age >18 years old

Exclusion Criteria:

1) Patients with VT due to a reversible cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed sustained scar-related VT who meet all of the following inclusion criteria will be eligible for enrollment
Sampling Method: Probability Sample
Enrollment: 2454 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Identification of the best sequence of treatments for a specific patient to optimize long-term outcomes | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Samuel, MPH, PhD, Principal Investigator — Montreal Heart Institute; John L Sapp, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (3):
- Canada (3):
  - Providence Health Care Society, Vancouver, British Columbia
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Montreal Heart Institute,, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No